CLINICAL TRIAL: NCT03899103
Title: Randomized Clinical Trial to Compare Efficacy and Safety of Repeated Courses of Rituximab to That of Maintenance Mycophenolate Mofetil Following Single Course of Rituximab in Maintaining Remission Over 24 Months Among Children With Steroid Dependent Nephrotic Syndrome
Brief Title: Compare Efficacy and Safety of Repeated Courses of Rituximab to That of Maintenance Mycophenolate Mofetil Following Single Course of Rituximab Among Children With Steroid Dependent Nephrotic Syndrome
Acronym: RITURNS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nilratan Sircar Medical College (Other Government)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Biswanath Basu, Associate Professor, Nilratan Sircar Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PednephroRCT/NMC/586
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Steroid-Dependent Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repeated Courses of Rituximab Only (Experimental): First course Course Rituximab at Randomization. Prophylactic 2nd and 3rd course rituximab re-administration will be done at 8 months and 16 months of follow-up if B cell count normalize.
  Interventions: Drug: Rituximab
- Rituximab and Mycophenolate Mofetil (Active Comparator): First course Course Rituximab at Randomization. Addition of Maintenance Mycophenolate Mofetil from 4 Month onwards.
  Interventions: Drug: Rituximab; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Rituximab — First course Course Rituximab at Randomization.
Drug: Mycophenolate Mofetil — Addition of Maintenance Mycophenolate Mofetil from 4 Month onwards
  Arms: Rituximab and Mycophenolate Mofetil

SUMMARY:
The aim of the RITURNS II study is to evaluate the efficacy and safety of Repeat courses of Rituximab to that of maintenance Mycophenolate Mofetil following single course of Rituximab in maintaining remission over 24 months among Children with Steroid Dependent Nephrotic Syndrome (SDNS).

DETAILED DESCRIPTION:
The vast majority of children with idiopathic nephrotic syndrome respond well to corticosteroid treatment. However, as many as 70% experience at least one relapse, and 30% develop a more complicated course with frequent relapses (FRNS) with or without steroid dependency (SDNS). Extended steroid exposure in these children often results in long-term complications. The management of patients with SDNS is challenging and expensive. Relapses may lead to serious complications, e.g. related to anasarca, hypertension, life threatening infections (peritonitis, pneumonia, meningitis), thrombosis and malnutrition. Repeated courses or even continuous steroid treatment lead to considerable medication related toxicity and morbidity.

The goal of treatment is to reduce the rate of relapses, the cumulative dose of corticosteroids, and the incidence of serious complications. Various prospective studies suggest that Rituximab, a B cell depleting monoclonal antibody, could be a safe and effective alternative to steroid or immunosuppressants to achieve and maintain remission in this population. Single rituximab infusion have been shown to be efficacious for 6 to 12 months and the side effect profile observed to date is very benign but after 6-8 months there was relapse due to regeneration of B-lymphocytes, hence for maintenance of remission MMF has been considered. In spite of good initial response, rituximab responders always remain prone to further relapse with regeneration of B lymphocytes, necessitating either repeat course of rituximab or addition of another steroid-sparing immunosuppressant. Reports suggest efficacy of rituximab may vary depending on disease pathology, clinical course, and simultaneous use of other immunosuppressants.

The aim of the RITURNS II study is to evaluate the efficacy and safety of Repeat courses of Rituximab to that of maintenance Mycophenolate Mofetil following single course of Rituximab in maintaining remission over 24 months among Children with Steroid Dependent Nephrotic Syndrome (SDNS).

ELIGIBILITY:
Inclusion Criteria

* Children between 3 and 16 years with SDNS.
* Minimal Change disease/ FSGS/MesPGN as per Kidney Biopsy report.
* Estimated glomerular filtration rate (eGFR) >80 ml/min per 1.73 m2 at study entry.
* Remission at study entry (Urine albumin nil or trace (or proteinuria <4 mg/m2/h) for 3 consecutive early morning specimens).
* Not received any steroid sparing agent previously.
* Parents willing to give informed written and audiovisual consent.
* Ability to swallow tablet.

Exclusion Criteria

* Known etiology (e.g., lupus erythematosus, IgA nephropathy, amyloidosis, malignancy, other secondary forms of NS).
* Patients with severe leukopenia (leukocytes <3.0× 1000 cells/mm3), severe anemia (haemoglobin <8.9 g/dl), thrombocytopenia (platelet <100.0 × 1000 cells/mm3) or deranged liver function tests (AST or ALT to >50 IU/L ) at enrolment.
* Known active chronic infection (tuberculosis, HIV, hepatitis B or C).
* Live vaccination within one month prior to screening.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the time to first relapse or death (whichever occurs first) till end of study (follow-up phase of 24 months) | 24 months

SECONDARY OUTCOMES:
Cumulative prednisolone requirement (mg/kg/yr) over the first 12 and 24 months, respectively. | 12 and 24 months
Number and severity of adverse events | 0-24 months
Number of relapses within months 0-24, 0-12 and 12-24, respectively | months 0-24, 0-12 and 12-24

CONTACTS AND LOCATIONS:
Locations (1):
- Nilratan Sircar Medical College and Hospital, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Chan EY, Yap DY, Colucci M, Ma AL, Parekh RS, Tullus K. Use of Rituximab in Childhood Idiopathic Nephrotic Syndrome. Clin J Am Soc Nephrol. 2023 Apr 1;18(4):533-548. doi: 10.2215/CJN.08570722. Epub 2023 Feb 22. PMID 36456193
- [Derived] Basu B, Preussler S, Sander A, Mahapatra TKS, Schaefer F. Randomized clinical trial to compare efficacy and safety of repeated courses of rituximab to single-course rituximab followed by maintenance mycophenolate-mofetil in children with steroid dependent nephrotic syndrome. BMC Nephrol. 2020 Nov 30;21(1):520. doi: 10.1186/s12882-020-02153-5. PMID 33256621